CLINICAL TRIAL: NCT00475059
Title: Performance of Cimetidine-corrected MDRD Equation in Renal Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Clément CAILLAUX, Centre Hospitalier Universitaire de Saint Etienne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0608090; 2006-005294-22
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Kidney Transplantation
Keywords: kidney transplantation; Glomerular filtration rate; inulin clearance; MDRD equation; cystatin C; cimetidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): patients who received cimétidine
  Interventions: Drug: cimetidine arrow

INTERVENTIONS:
Drug: cimetidine arrow — patients who received cimétidine

SUMMARY:
Among the different creatinine-based GFR predicting equations, the MDRD equation gives the best prediction in renal transplantation but does not provide the level of accuracy usually seen in renal patients with native kidneys.

Blocking the tubular secretion of creatinine with an oral administration of cimetidine is likely to make creatinine a more accurate marker of GFR.

We will test the hypothesis that the accuracy of the MDRD equation will be improved in renal transplant patients by incorporating into the equation a cimetidine-corrected serum creatinine value.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplantation > 1 year
* Patient with immunosuppressant treatment of TACROLIMUS (PROGRAF)
* Creatinine clearance > 30 ml/min/1,73m2 within 3 months before inclusion
* Written informed consent
* Patient affiliated to social insurance

Exclusion Criteria:

* Unstable renal function defined by serum creatinine (J0) > 25% serum creatinine realised in 3 months
* Treatment: Bactrim, Fansidar, Cimetidine arrow within the week before inclusion
* Contraindication listed in the labeling of Cimetidine arrow
* Last residual rate of Tacrolimus > 12 ng/ml.
* Treatment : carvedilol, phenytoïn (interaction with cimetidine)
* Serious hepatic insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
performance of inulin clearance and MDRD with or no block of secretion renal tubule with cimetidine | two days

SECONDARY OUTCOMES:
Performance of different prediction equations for estimating renal function with or no block of secretion renal tubule with cimetidine : - Walser equation - Nankivell equation - Cockcroft and Gault equation | two days
comparison between inulin clearance and cystatin C | two days

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Mariat, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Nephrology unit, CHU Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Mariat C, Alamartine E, Afiani A, Thibaudin L, Laurent B, Berthoux P, De Filippis JP, Thibaudin D, Mayor B, Elessawy AB, Berthoux F. Predicting glomerular filtration rate in kidney transplantation: are the K/DOQI guidelines applicable? Am J Transplant. 2005 Nov;5(11):2698-703. doi: 10.1111/j.1600-6143.2005.01070.x. PMID 16212629
- [Background] Mariat C, Alamartine E, Barthelemy JC, De Filippis JP, Thibaudin D, Berthoux P, Laurent B, Thibaudin L, Berthoux F. Assessing renal graft function in clinical trials: can tests predicting glomerular filtration rate substitute for a reference method? Kidney Int. 2004 Jan;65(1):289-97. doi: 10.1111/j.1523-1755.2004.00350.x. PMID 14675062
- [Background] Gaspari F, Ferrari S, Stucchi N, Centemeri E, Carrara F, Pellegrino M, Gherardi G, Gotti E, Segoloni G, Salvadori M, Rigotti P, Valente U, Donati D, Sandrini S, Sparacino V, Remuzzi G, Perico N; MY.S.S. Study Investigators. Performance of different prediction equations for estimating renal function in kidney transplantation. Am J Transplant. 2004 Nov;4(11):1826-35. doi: 10.1111/j.1600-6143.2004.00579.x. PMID 15476483
- [Background] Bosma RJ, Doorenbos CR, Stegeman CA, van der Heide JJ, Navis G. Predictive performance of renal function equations in renal transplant recipients: an analysis of patient factors in bias. Am J Transplant. 2005 Sep;5(9):2193-203. doi: 10.1111/j.1600-6143.2005.00982.x. PMID 16095498
- [Background] Poge U, Gerhardt T, Palmedo H, Klehr HU, Sauerbruch T, Woitas RP. MDRD equations for estimation of GFR in renal transplant recipients. Am J Transplant. 2005 Jun;5(6):1306-11. doi: 10.1111/j.1600-6143.2005.00861.x. PMID 15888034
- [Background] Poggio ED, Wang X, Weinstein DM, Issa N, Dennis VW, Braun WE, Hall PM. Assessing glomerular filtration rate by estimation equations in kidney transplant recipients. Am J Transplant. 2006 Jan;6(1):100-8. doi: 10.1111/j.1600-6143.2005.01140.x. PMID 16433763
- [Background] Kemperman FA, Surachno J, Krediet RT, Arisz L. Cimetidine improves prediction of the glomerular filtration rate by the Cockcroft-Gault formula in renal transplant recipients. Transplantation. 2002 Mar 15;73(5):770-4. doi: 10.1097/00007890-200203150-00020. PMID 11907426
- [Background] Nankivell BJ, Gruenewald SM, Allen RD, Chapman JR. Predicting glomerular filtration rate after kidney transplantation. Transplantation. 1995 Jun 27;59(12):1683-9. doi: 10.1097/00007890-199506270-00007. PMID 7604438
- [Background] Myara I, Lahiani F, Cosson C, Duboust A, Moatti N. Estimated creatinine clearance by the formula of Gault and Cockcroft in renal transplantation. Nephron. 1989;51(3):426-7. doi: 10.1159/000185340. No abstract available. PMID 2645534
- [Background] Goerdt PJ, Heim-Duthoy KL, Macres M, Swan SK. Predictive performance of renal function estimate equations in renal allografts. Br J Clin Pharmacol. 1997 Sep;44(3):261-5. doi: 10.1046/j.1365-2125.1997.t01-1-00567.x. PMID 9296320
- [Background] Perico N, Gaspari F, Remuzzi G. Assessing renal function by GFR prediction equations in kidney transplantation. Am J Transplant. 2005 Jun;5(6):1175-6. doi: 10.1111/j.1600-6143.2005.00939.x. No abstract available. PMID 15888019
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Froissart M, Rossert J, Jacquot C, Paillard M, Houillier P. Predictive performance of the modification of diet in renal disease and Cockcroft-Gault equations for estimating renal function. J Am Soc Nephrol. 2005 Mar;16(3):763-73. doi: 10.1681/ASN.2004070549. Epub 2005 Jan 19. PMID 15659562
- [Background] Poggio ED, Wang X, Greene T, Van Lente F, Hall PM. Performance of the modification of diet in renal disease and Cockcroft-Gault equations in the estimation of GFR in health and in chronic kidney disease. J Am Soc Nephrol. 2005 Feb;16(2):459-66. doi: 10.1681/ASN.2004060447. Epub 2004 Dec 22. PMID 15615823
- [Background] White C, Akbari A, Hussain N, Dinh L, Filler G, Lepage N, Knoll GA. Estimating glomerular filtration rate in kidney transplantation: a comparison between serum creatinine and cystatin C-based methods. J Am Soc Nephrol. 2005 Dec;16(12):3763-70. doi: 10.1681/ASN.2005050512. Epub 2005 Oct 19. PMID 16236805
- [Background] Lemahieu WP, Maes BD, Verbeke K, Vanrenterghem Y. Impact of gastric acid suppressants on cytochrome P450 3A4 and P-glycoprotein: consequences for FK506 assimilation. Kidney Int. 2005 Mar;67(3):1152-60. doi: 10.1111/j.1523-1755.2005.00182.x. PMID 15698457